CLINICAL TRIAL: NCT02488798
Title: The Role of Office Hysteroscopy and Endometrial Power Doppler Using the International Endometrial Tumor Analysis Group Classification in the Evaluation of Postmenopausal Bleeding
Brief Title: Office Hysteroscopy and 3D Power Doppler Vaginal Ultrasound in Assessment of Postmenopausal Bleeding
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yasmin Ahmed Bassiouny, Dr, Cairo University
Other Study IDs: 62014
Record Dates: First submitted 2015-06-30; First posted 2015-07-02 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2015-06

CONDITIONS: Postmenopausal Bleeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sample from the uterine endometrium for histopathological analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- postmenopausal bleeding group: 100 women with postmenopausal bleeding undergoing 2D greyscale vaginal ultrasound and 3D Endometrial power Doppler and the features were classified using six different vascular patterns described by IETA group including the following patterns; single dominant vessel without branching, with branching, multiple vessels with focal origin, with multifocal origin at the myometrium-endometrium junction, scattered vessels or circular flow (Kucur et al., 2013 ).
  All patients then had Office hysteroscopy carried out in the outpatient clinic using vaginoscopic approach (Cooper et al., 2010). With endometrial samples from lesions or from the cavity for histopathological analysis.
  Interventions: Procedure: 2D grey scale vaginal ultrasound; Procedure: 3D power Doppler vaginal ultrasound; Procedure: Office hysteroscopy

INTERVENTIONS:
Procedure: 2D grey scale vaginal ultrasound — To assess the endometrial thickness and echogenicity (whether the endometrium is uniform or non-uniform).
Procedure: 3D power Doppler vaginal ultrasound — To assess the endometrium using the IETA group criteria.
Procedure: Office hysteroscopy — using the vaginoscopic approach to assess the uterine cavity and take sample.

SUMMARY:
100 patients with postmenopausal bleeding were assessed with 2D vaginal ultrasound and 3D power Doppler ultrasound using the international endometrial tumor analysis group and office hysteroscopy with taking samples for histopathological analysis.

DETAILED DESCRIPTION:
The aim was to compare the efficiency of the upper mentioned interventions in diagnosing the cause of postmenopausal bleeding.

ELIGIBILITY:
Inclusion Criteria:

* 100 patients complaining of postmenopausal bleeding. Postmenopausal bleeding was defined as vaginal bleeding that occurred after at least 12 months of amenorrhea.

Exclusion Criteria:

* Exclusion criteria included any history of hormone administration in the last 6 months, any medical condition that might cause abnormal uterine bleeding like coagulation disorders, hypertension, cardiac disease, thyroid disorders or hepatic condition.

Ages: 47 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with postmenopausal bleeding
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Efficacy of 3D power Doppler ultrasound with the IETA group criteria in diagnosing the cause of postmenopausal bleeding | 1 week
  Efficacy of 3D power Doppler ultrasound with the IETA group criteria in diagnosing the cause of postmenopausal bleeding